CLINICAL TRIAL: NCT06040775
Title: Evaluation of Theta Burst Transcranial Magnetic Stimulation as an Adjunct to Standard Therapy in Improving Core Function Deficits in Children 5-15 Year Age With Autism Spectrum Disorder - a Randomized, Double Blind, Sham Controlled Trial
Brief Title: Evaluation of Theta Burst Transcranial Magnetic Stimulation in Children With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TBS-ASD
Record Dates: First submitted 2023-07-03; First posted 2023-09-18 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Theta burst transcranial magnetic stimulation arm (Experimental): Theta burst transcranial magnetic stimulation with Applied Behaviour Analysis
  Interventions: Device: Theta Burst Transcranial magnetic Stimulation using real MCF-B65 coil
- Sham arm (Sham Comparator): Sham transcranial magnetic stimulation with Applied Behaviour Analysis
  Interventions: Device: Sham magnetic stimulation using sham MCF-B65 coil

INTERVENTIONS:
Device: Theta Burst Transcranial magnetic Stimulation using real MCF-B65 coil — Site of stimulation will be predetermined at Dorsolateral prefrontal cortex of non-dominant side using the BeamF3 method.1 burst will be - 3 pulses at 50 Hz, burst will be set at 5Hz i.e. interburst interval 200ms .
  At100% of resting motor threshold of dominant side - 5 trains (each 40sec on and 20 sec off) will be given at each session with a pause of 1 minute in between 2 trains Standard therapy with Applied Behavior Analysis and sensory integration would continue
  Other Names: Applied Behavioral Analysis
  Arms: Theta burst transcranial magnetic stimulation arm
Device: Sham magnetic stimulation using sham MCF-B65 coil — Similar set parameters using a sham coil which simulates sound and tactile effect of real coil but no electromagnetic induction is produced.
  Standard therapy with Applied Behavior Analysis and sensory integration would continue
  Other Names: Applied Behavioral Analysis
  Arms: Sham arm

SUMMARY:
The goal of this clinical trial is to evaluate Theta Burst Transcranial Magnetic Stimulation as an adjunct to standard therapy in improving core function deficits in children 5-15 year age with Autism Spectrum disorder. The main question it aims to answer is whether Theta burst Transcranial Magnetic Stimulation would improve core function deficit in children age 5 - 15 years with Autism Spectrum Disorder as an adjunct to standard therapy. Participants will receive patterned transcranial magnetic stimulation- theta burst stimulation for consecutive 7 days with standard therapy and the comparison group would receive standard therapy alone. Outcome in the form of change in obsessive, repetitive behavior would be measured at 1 month from end of therapy

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder with varying degrees of severity and symptoms with core deficits in social communication and interaction and repetitive behavior with restricted interests and activities -American Psychiatric Association, 2013. Diagnosis requires fulfilment of DSM V criterion for Autism Spectrum Disorder. ASD is a lifelong disorder with onset in early developmental period and most patients remain severely impaired in terms of psychosocial functioning throughout their adult lives.

Need for exploration of newer treatment modalities - Currently there is no definitive treatment of Autism and for now the management strategies include - Applied Behavioral Analysis (ABA), sensory integration, and structured teaching targeting core deficits which are time taking process and labor intensive from both the caregiver and the provider's perspective. Pharmacotherapy is effective for targeting associated comorbidities like irritability, aggression, destructive behavior or hyperactivity and had the added disadvantage of side effects like sedation. For Complementary and Alternative Medicine strategies, proof of efficacy has not been unestablished for many. In this context Transcranial Magnetic Stimulation, TMS may prove to be a good non-invasive neuromodulation technique and could be an effective tool in the treatment of ASD core manifestations.

Transcranial Magnetic Stimulation (TMS) is a non-invasive neuromodulation technique. It uses electromagnetic induction to generate transient, localized electrical fields in the brain cortex, causes depolarization and firing of local neurons. Acute effects of TMS include phasic activation of neural circuits and prolonged effects of TMS include alteration in Neuroplasticity by change in synaptic efficacy, leading to long term potentiation or long-term depression, this occurs via alteration in neurotropic factor, modulation of cortical excitability, modulation of functional connectivity. The current study aims to explore role of patterned TMS known as Theta Burst Stimulation (TBS)- in which pulses are applied in bursts of three, frequency of 50 Hz and an inter-burst interval of 200 milli seconds. TBS is a patterned form of repetitive transcranial magnetic stimulation (rTMS) modelled after endogenous hippocampal discharge patterns and has been shown to be more efficient than standard rTMS in modulating cortical excitability. The potential advantages of TBS over rTMS, particularly for children with ASD include shorter overall stimulation duration (5minutes in TBS). Also, TBS could be better tolerated overall and perhaps even safer than standard rTMS as sub threshold intensities are given for shorter periods. Effects of TBS on synaptic plasticity occur much more rapidly than with traditional repetitive TMS protocols. It is also less noisy due to lower amplitudes used which may reduce hyper sensory stimulation and may be one of the reasons why TBS could be better tolerated in children with ASD There seems to be converging in implication of role of dorsolateral prefrontal cortex in pathophysiology and aberrant neural circuitry of children with ASD. This study aims to study the effect of TBS as an adjunct to the ongoing standard therapy on core deficits in autism as measured by CY-BOCS - Children's Yale-Brown Obsessive Compulsive Scale, RBS-R - Repetitive Behavior Scale- Revised, social behavior change as measured by SRS-2 - Social Responsiveness Scale- version 2 and overall autistic traits using CARS-2 - Childhood Autism Rating Scale- version 2 at 1 month and 3 month from end of TBS sessions. It also aims to measure parent reported quality of life and adverse event rates participants. Change in cognitive function using Wisconsin card sorting and time to stroop will be used in participants with IQ>70.

ELIGIBILITY:
Inclusion Criteria:

1. 5 to 15 year age.
2. Fulfills DSM-V diagnosis of autism spectrum disorder (ASD)

Exclusion Criteria:

1. Secondary causes of autism

   * Global developmental delay, hearing or vision abnormality
   * Structural brain abnormalities on imaging
   * Genetic or syndromic associations- Down's/Fragile X/Rett's syndrome
2. Children on unstable drug regimen- (antipsychotics or anti epileptics) for last 1 months will be excluded
3. Neurological or psychiatric disorder other than comorbid disorders of ASD
4. Uncontrolled epilepsy as defined by seizure frequency >1/month for preceding 3 months (including diagnosed patients with CSWS/LKS)
5. Severe concurrent illness or disease or unstable medical conditions like pneumonia
6. Any contraindications for TMS Implanted electronic device and non-removable metallic objects near coil e.g., pacemaker, cochlear implant Presence of ferromagnetic metal in the head outside the mouth On medication lowering seizure threshold

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in core function deficit in obsessive and repetitive behavior between intervention and control arm | 4 weeks +/- 3 days from end of therapy
  Difference in mean change in total Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) and Repetitive Behaviors Scale - Revised (RBS-R) score between intervention and control group
  CYBOCS- Clinician-report questionnaire, 70 questions, Each on scale of of 0-4, Maximum score -280, minimum score- 0. Higher scores suggest mores severe symptoms RBS-R - Self report/caregiver, 44-item, Each on scale of of 0-4, Maximum score -176, minimum- 0. Higher scores suggest mores severe symptoms

SECONDARY OUTCOMES:
Change in core function deficit in social behavior and overall autism score between intervention and control arm | 4 weeks +/- 3 days from end of therapy
  Difference in mean change in total Social Responsiveness Scale, Second Edition (SRS-2) and Childhood Autism Rating Scale, Second Edition (CARS-2) scores between intervention and control group
  SRS-2- Parent or teacher questionnaire (65 items on a 4- point Likert scale), Five domain scores ("Treatment Subscales"), Expressed as a raw score or a T-scores. Higher scores more severe social impairment CARS-2 -15 item scale, 1-4 in key areas related to autism diagnosis. For under 12 years of age, scores of 30 or above are indicative of autism and for students 12 years and older, scores of 28 or above are considered to be indicative of autism.
Change in core function deficit in social behavior and overall autism score between intervention and control arm | 12 weeks +/- 7 days from end of therapy
  Difference in mean change in total CY-BOCS, RBS-R, SRS-2, CARS-2 scores between intervention and control group CYBOCS- Clinician-report questionnaire, 70 questions, Each on scale of of 0-4, Maximum score -280, minimum score- 0. Higher scores suggest mores severe symptoms RBS-R - Self report/caregiver, 44-item, Each on scale of of 0-4, Maximum score -176, minimum- 0. Higher scores suggest mores severe symptoms SRS-2- Parent or teacher questionnaire (65 items on a 4- point Likert scale), Five domain scores ("Treatment Subscales"), Expressed as a raw score or a T-scores. Higher scores more severe social impairment CARS-2 -15 item scale, 1-4 in key areas related to autism diagnosis. For under 12 years of age, scores of 30 or above are indicative of autism and for students 12 years and older, scores of 28 or above are considered to be indicative of autism.
Change in parent reported quality of life as assessed by PedsQL score between intervention and control arm | 4 weeks +/- 3 days from end of therapy and 12 weeks +/- 7 days from end of therapy
  Difference in mean change in total Pediatric Quality of Life Inventory (PedsQL) score between intervention and control group
Describe Adverse events noted in intervention and control arm | 4 weeks +/- 3 days from end of therapy
  Adverse event rate defined as ratio of sessions with adverse events divided by total sessions
  Adverse event will be defines as- positive increase in any of the ROS (review of systems) criteria compared to pre therapy (which will be filled at end of each therapy session)
To describe effect of TBS in clinical tests for executive function using Wisconsin Card Sorting Test (in study population with IQ>70) | at first visit, at 4 weeks +/- 3 days from end of therapy and at 12 weeks from end of therapy
  Wisconsin Card Sorting Test- Mean of change in total error score will be calculated for intervention and control arms
To describe effect of TBS in clinical tests for executive function using Stroop test time(in study population with IQ>70) | at first visit, at 4 weeks +/- 3 days from end of therapy and at 12 weeks from end of therapy
  Stroop test time- Total time to complete 3 paged stroop test (in seconds) will be compared or intervention and control arms

CONTACTS AND LOCATIONS:
Overall Officials: Sheffali Gulati, Principal Investigator — All India Institute of Medical Sciences

IPD SHARING:
Plan to Share IPD: No